CLINICAL TRIAL: NCT03887039
Title: Oral Findings In A Group of Egyptian Children With Attention Deficit Hyperactivity Disorder: A Cross-Sectional Study
Brief Title: Oral Findings In A Group of Egyptian Children With Attention Deficit Hyperactivity Disorder
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Gaber Hussien, Principal investigator, Cairo University
Other Study IDs: 14422016496994
Record Dates: First submitted 2019-03-19; First posted 2019-03-22 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-03

CONDITIONS: Oral Manifestations
Keywords: oral findings; oral characteristics; oral health; caries; oral habits; dental trauma; ADHD; children
MeSH Terms: conditions — Oral Manifestations; Attention Deficit Disorder with Hyperactivity | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ADHD group: clinical examination
  Interventions: Other: clinical examination
- normal group: clinical examination
  Interventions: Other: clinical examination

INTERVENTIONS:
Other: clinical examination — clinical examination for all the oral findings

SUMMARY:
Attention-deficit/hyperactivity disorder is the most common childhood neuro-developmental disorder that is characterized by inattention, hyperactivity, and impulsivity. These symptoms last till adulthood in 65% of cases. ADHD has been reported to have a worldwide prevalence of 5.3% and it is more common in boys than in girls (Ghanizadeh 2008; Serra-Negra et al. 2012 and Shooshtari et al. 2013) The symptoms of ADHD are generally treated through behavioral therapy, with or without pharmacological intervention. Medications prescribed are commonly divided into stimulant or non-stimulant drugs. The stimulant medications (such as methylphenidate and amphetamines) have been implicated in adverse oral effects, such as xerostomia and gingival enlargement. The current evidence is controversial regarding the severity and prevalence of dental caries, dental trauma, periodontal diseases, oral habits and tooth wear among patients with ADHD (Chau et al. 2017).

In the Arab world, few studies have been published on ADHD. Accordingly, in the Arab society and Egypt there are limited data regarding the oral findings of children with ADHD. Owing to the sparsity of these data, this study will be conducted to evaluate different oral characteristics of Egyptian children with ADHD.

DETAILED DESCRIPTION:
Due to lack of published studies about the oral findings of Egyptian Children with ADHD, this study will be conducted to cover this point.

ELIGIBILITY:
Inclusion Criteria:

* - Egyptian children 3-6 years old diagnosed with ADHD.
* Patients taking medications for the treatment of ADHD or not.
* Both male and female patients will be included.

Control Group:

A matched group of healthy children aged 3-6 years old.

Exclusion Criteria:

* - Non-Egyptian children.
* Patients having systemic disorders, such as cerebral palsy or Down's syndrome.
* Patients complaining from any systemic disease

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients referred from Abu El-Reesh and El-Demerdash children hospitals, diagnosed with ADHD.
  Control group: A matched group of patients attending at Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Cairo University.
  Patients will be included in the study according to the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
oral habits | 6 months
  clinical examination yes/no

SECONDARY OUTCOMES:
DMFT caries index | 6 months
  DMFT D=dacayed M=missed due to caries F=filled T=tooth score 0-20 for primary teeth0 is the best / 20 is the worst
dental trauma | 6 months
  clinical examination yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Sara G Hussien, BSc, Principal Investigator — Resident at pediatric Dentistry and Dental Public Health Department; Randa Y Abdel Gawad, PhD, Study Director — Associate professor at pediatric Dentistry and Dental Public Health Department

IPD SHARING:
Plan to Share IPD: Yes